CLINICAL TRIAL: NCT01772069
Title: Health-Related Quality of Life in Patients With Systemic Lupus Erythematosus:Focusing on Fibromyalgia
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jun-Ki Min, Professor, The Catholic University of Korea
Other Study IDs: HC12QIMI0020
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Quality of Life
Keywords: systemic lupus erythematosus, disease activity, sleep, quality of life
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Systemic lupus erythematosus (SLE) patients show a high prevalence of fibromyalgia though rates vary considerably from one study to another (from 8.2% to 45%). Although fibromyalgia can bring out the disability in daily life, the majority of previous reports only ascertained no significant association between the presence of fibromyalgia and the severity of SLE.

It is necessary to make unremitting effort to reduce the mortality and life-threatening disease flare-up due to SLE disease itself. Additionally, we think that physicians need to pay more attention to improve health-related quality of life (HRQoL) in the patients with SLE. HRQoL could be influenced by various factors such as depression, fibromyalgia, disease duration, disease activity and etc. To improve the HRQoL in SLE patients, it might be the clinically important and constructive theme to investigate that which is the most important factor among the fibromyalgia, depression, sleep quality, SLE activity and SLE duration.

The objective of this study is to evaluate the degree of contribution of fibromyalgia for reduced HRQoL and to identify the status of managing fibromyalgia in Korean patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Woman between 30 and 60 years of age, inclusive
2. Have a diagnosis of Systemic lupus erythematosus according to the 1997 updated American college of Rheumatology criteria for classification of systemic lupus erythematosus

Exclusion Criteria:

1. Patients were excluded if they had had a history of head injury that led to unconsciousness
2. Have unstable disease necessitating an increase in prednisone dose or the addition of another immunosuppressive medication
3. Have a current malignancy
4. Have a history of or current evidence of substance abuse (drug or alcohol) problem within the previous 2 years

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Patients : 150 women age 30 to 60 years with SLE
  * Control subjects : age, sex matched control subject (150 subjects)
  * Patients : First visit and second visit after an interval of six months
  * Control subjects : baseline only
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
EuroQoL (EQ-5D) | 1 year